CLINICAL TRIAL: NCT01666561
Title: The Effect of Oat Based Breakfast Cereals on Satiety and Food Intake.
Acronym: Quaker A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frank Greenway (Other)
Collaborators: PepsiCo Global R&D (Industry); Quaker Oats Company (Industry)
Responsible Party: Sponsor-Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Organization: Pennington Biomedical Research Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PBRC 12029 (Period 1)
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Food Intake; Satiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Breakfast Test Cereal 1, Oat based (Experimental): Test cereal 1, Oat based breakfast cereal- you will be randomly presented with a breakfast consisting of either:
  Oat-based breakfast cereal with lactose-free, fat-free milk to drink or ready-to-eat cereal in lactose-free, fat -free milk with water to drink. Then you will complete a visual analog scale at 30, 60, 120. 180, and 240 minutes following the start of breakfast meal.
  Interventions: Other: Breakfast Test Cereal 1, Oat based; Other: Breakfast Test Cereal 2, Oat-based; Other: Ready-to-eat cereal
- Breakfast Test Cereal 2, Oat-based (Experimental): Test Cereal 2, Oat-based breakfast cereal. You will be randomly presented with a breakfast consisting of either:
  Oat-based breakfast cereal with lactose-free, fat-free milk to drink or ready-to-eat oat brand cereal in lactose-free, fat -free milk with water to drink. Then you will complete a visual analog scale at 30, 60, 120. 180, and 240 minutes following the start of breakfast meal.
  Interventions: Other: Breakfast Test Cereal 1, Oat based; Other: Breakfast Test Cereal 2, Oat-based; Other: Ready-to-eat cereal
- Ready-to-eat cereal (Experimental): Ready-to-eat cereal, Oat based breakfast cereal- you will be randomly presented with a breakfast consisting of either:
  one Oat-based breakfast cereal with lactose-free, fat-free milk to drink or ready-to-eat cereal in lactose-free, fat -free milk with water to drink. Then you will complete a visual analog scale at 30, 60, 120. 180, and 240 minutes following the start of breakfast meal.
  Interventions: Other: Breakfast Test Cereal 1, Oat based; Other: Breakfast Test Cereal 2, Oat-based; Other: Ready-to-eat cereal

INTERVENTIONS:
Other: Breakfast Test Cereal 1, Oat based — The study design is a crossover trial with each subject receiving one of the cereals in each of three visits separated by at least a week will be enrolled to investigate the satiety impact of three breakfast cereals: (a) one serving of oat based breakfast cereal 1.
Other: Breakfast Test Cereal 2, Oat-based — The study design is a crossover trial with each subject receiving one of the cereals in each of three visits separated by at least a week will be enrolled to investigate the satiety impact of three breakfast cereals: (b) an equicaloric amount of Oat based breakfast cereal 2.
Other: Ready-to-eat cereal — The study design is a crossover trial with each subject receiving one of the cereals in each of three visits separated by at least a week will be enrolled to investigate the satiety impact of three breakfast cereals: (c) an equicaloric amount of the ready-to-eat cold cereal.

SUMMARY:
To test the hypothesis that two 40 gm serving of Oat-based breakfast cereals compared to an equicaloric amount of a ready-to-eat Oat-based breakfast cereal will give greater satiety over the 4 hour period following breakfast.

DETAILED DESCRIPTION:
The subjects will be randomly assigned to one of these three breakfasts and then given a Visual analogue scales of hunger and satiety which will be completed at baseline, 30, 60, 120, 180, and 240 minutes. Subjects will return on 2 other days separated by at least a week to repeat the breakfast test.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and are healthy.
* Taking no regular medications other than birth control or hormone replacement therapy.
* Are willing to use an effective method of birth control if you are capable of bearing children. Acceptable methods include abstinence, barrier methods, intrauterine devices, and hormonal methods of contraception.

Exclusion Criteria:

* Are a woman who is pregnant or nursing a baby.
* Have gained or lost 8.8 pounds or more in the last 3 months.
* Have diabetes or a fasting blood sugar over 126 mg/dL.
* Have a score of 14 or greater on the restraint scale of the 3-factor eating questionnaire (a questionnaire which will be given to you by the study staff).
* Are allergic to oats, lactose-free milk, Honey Nut Cheerios or oatmeal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Satiety Impact | up to day 3
  Breakfast containing of oat-based breakfast cereal will cause people to feel more satiated compared to a breakfast containing of ready-to-eat oat-based breakfast cereal. Appetite and satiety will be measured with a Visual Analog Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States